CLINICAL TRIAL: NCT03130023
Title: The Relationship Between Oxygen Reserve Index and PaO2 in Children
Brief Title: The Relationship Between Oxygen Reserve Index and PaO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PED ORI
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Children; Congenital Heart Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test group (Experimental): All subjects will be enrolled in the test group and will receive Pulse Oximeter with ORI.
  Interventions: Device: Pulse Oximeter with ORI

INTERVENTIONS:
Device: Pulse Oximeter with ORI — Pulse oximeter that measure Oxygen Reserve Index

SUMMARY:
Oxygen Reserve Index (ORI) is a new parameter for noninvasive monitoring of oxygen reserve using oximetry sensor. In this study, the investigators evaluate the correlation between ORI and the partial pressure of arterial blood oxygen (PaO2) in children.

ELIGIBILITY:
Inclusion Criteria:

* Age below 7 years
* Written informed consent
* Undergoing cardiac surgery

Exclusion Criteria:

* Presence of cyanotic heart disease

Max Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
correlation coefficient between ORI and PaO2 | through study completion, an average of 5 hours
  correlation coefficient between ORI and PaO2

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim JT, Park JB, Ji SH, Jang YE, Kim EH, Kim HS, Lee JH. Dynamics of Oxygen Reserve Index and Arterial Oxygen Partial Pressure in Children: A Prospective Observational Study. Paediatr Anaesth. 2025 Oct;35(10):810-815. doi: 10.1111/pan.70014. Epub 2025 Jul 21. PMID 40686277